CLINICAL TRIAL: NCT04214067
Title: A Phase III Randomized Trial of Radiation +/- Pembrolizumab (MK-3475) for Newly Diagnosed Early Stage High Intermediate Risk Mismatch Repair Deficient (dMMR) Endometrioid Endometrial Cancer
Brief Title: Testing the Addition of the Immunotherapy Drug, Pembrolizumab, to the Usual Radiation Treatment for Newly Diagnosed Early Stage High Intermediate Risk Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-08602; NCI-2019-08602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY020 (Other: NRG Oncology); NRG-GY020 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Endometrioid Adenocarcinoma; Stage I Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8; Stage II Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8
MeSH Terms: conditions — Carcinosarcoma | interventions — Specimen Handling; Brachytherapy; Congresses as Topic; Radiation; Magnetic Resonance Spectroscopy; pembrolizumab; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (EBRT, brachytherapy) (Active Comparator): Patients undergo pelvic EBRT daily for 5-6 weeks and vaginal brachytherapy completed within 7 days after completion of EBRT in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and CT scans, MRI scans, or x-ray imaging throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Radiation: Brachytherapy; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: X-Ray Imaging
- Arm II (EBRT, brachytherapy, pembrolizumab) (Experimental): Patients undergo EBRT and brachytherapy as in Arm I. Within 7 days prior to the start of radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 6 weeks for up to 1 year (9 cycles) in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and CT scans, MRI scans, or x-ray imaging throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Radiation: Brachytherapy; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Brachytherapy — Undergo vaginal brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm II (EBRT, brachytherapy, pembrolizumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: X-Ray Imaging — Undergo x-rays
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase III trial compares whether the addition of pembrolizumab to radiation therapy is more effective than radiation therapy alone in reducing the risk of cancer coming back (recurrence) in patients with newly diagnosed stage I-II endometrial cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. The addition of pembrolizumab to radiation treatment may be more effective than radiation treatment alone in reducing cancer recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the 3-year recurrence-free survival of women with high intermediate risk (HIR) stage I/II mismatch repair deficient (dMMR) endometrioid endometrial cancer treated with radiation and pembrolizumab (MK-3475) versus radiation alone.

SECONDARY OBJECTIVES:

I. To describe the safety and tolerability of concurrent pembrolizumab (MK-3475) and radiation compared to radiation alone in patients with MMR deficient high intermediate risk endometrial cancer (HIR EC).

II. To describe the recurrence patterns in each group. III. To measure recurrence free survival at 5 years in each group. IV. To estimate disease specific overall survival in each group. V. To determine whether the addition of pembrolizumab (MK-3475) to radiation, compared with radiation alone is associated with decreased quality of life at 6- and 24-weeks, as measured with the Functional Assessment of Cancer Therapy (FACT)-Endometrial (En) Trial Outcome Index (TOI), increased gastrointestinal (GI) symptoms as measured with the GI subscale, and increased fatigue as measured with the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue scale (short form).

VI. To validate the Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM) subscale, which assesses in cancer patients on immunotherapy.

VII. To evaluate the ability of ctDNA to predict outcomes in the experimental and control groups.

CORRELATIVE/TERTIARY OBJECTIVES:

I. To explore the baseline tumor genetic and microenvironment parameters predictive of clinical benefit or resistance to immunotherapy.

II. To determine whether the addition of pembrolizumab (MK-3475) to radiation, compared with radiation alone, is associated with decreased quality of life as measured with the Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM subscale) and more self-reported bother from side effects as measured with a single item GP5 "I am bothered by side effects," a question from the FACT-En TOI.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo pelvic external beam radiation therapy (EBRT) daily for 5-6 weeks and vaginal brachytherapy completed within 7 days after completion of EBRT in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo EBRT and brachytherapy as in Arm I. Within 7 days prior to the start of radiation therapy, patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment with pembrolizumab repeats every 6 weeks for up to 1 year (9 cycles) in the absence of disease progression or unacceptable toxicity.

Patients in both arms also undergo collection of blood samples and computed tomography (CT) scans, magnetic resonance imaging (MRI) scans, or x-ray imaging throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have:

  * Stage I endometrioid endometrial cancer and a combination of age and risk factors as listed below:

    * Age >= 70 and 1 or more risk factors
    * Age 50 - < 70 and 2 or more risk factors
    * Age < 50 and 3 risk factors

      * Risk factors:

        * Myometrial invasion >= 50%
        * Lymphovascular space invasion
        * Grade 2 or 3 OR
  * Stage II endometrioid endometrial cancer

    * Note: Patients with isolated tumor cells in sentinel lymph nodes are eligible (considered N0i) as long as there is no evidence of micro- or macro-metastases in any lymph nodes
* CT or MRI abdomen or pelvis and either chest X-ray or CT chest demonstrating no evidence of disease outside of the uterus. Imaging can be performed pre-operatively or post-operatively. CT with contrast is the preferred modality. Positron emission tomography (PET)/CT is NOT to be used for any disease assessment or reassessment unless there is documentation that PET/CT is of diagnostic quality equal to CT with contrast
* Patients must have deficient mismatch repair as demonstrated by lack of expression of at least one mismatch repair protein by immunohistochemistry (IHC) and/or evidence of microsatellite instability (MSI) high. The institutional pathology report documenting MMR deficiency must be submitted
* Patients must have undergone surgical staging with at least hysterectomy, removal of cervix, bilateral (if both are present) salpingo-oophorectomy, and either sentinel lymph node assessment or complete pelvic +/- aortic lymphadenectomy. Secondary staging is allowed to determine stage. Patients with isolated tumor cells in sentinel lymph nodes are eligible (considered N0i) as long as there is no evidence of micro- or macro-metastases in any lymph nodes
* Patients must have received no prior therapy for endometrial cancer, including hormonal therapy, chemotherapy, targeted therapy, immunotherapy or radiation therapy
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Platelets >= 100,000/mcl (within 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500/mcl (within 14 days prior to registration)
* Creatinine =< 1.5 x laboratory upper limit of normal (ULN) (within 14 days prior to registration)
* Bilirubin =< 1.5 x ULN (within 14 days prior to registration) (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 14 days prior to registration)
* Thyroid stimulating hormone (TSH) within normal limits (TSH < ULN allowed in euthyroid patients on thyroid replacement therapy)
* Patients must be registered between 1 and 8 weeks after initial (staging) surgery performed for the combined purpose of diagnosis and staging
* Human immunodeficiency virus (HIV) testing is not required by protocol unless clinically indicated. Known HIV positive patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Patients who are currently participating and receiving cancer-directed study therapy for endometrial cancer or have participated in a study of an investigational agent and received cancer-directed study therapy for endometrial cancer within 4 weeks prior to registration
* Patients who have received prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapeutic antibody or other similar agents
* Patients who have a history of a severe hypersensitivity reaction to monoclonal antibody or MK-3475 (pembrolizumab) and/or its excipients
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. This includes, but is not limited to, patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including type I diabetes mellitus, thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients with a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registration:

  * Patients who have received steroids as CT scan contrast premedication may be enrolled
  * The use of inhaled or topical corticosteroids is allowed
  * The use of mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
  * The use of physiologic doses of corticosteroids may be approved after consultation with the study chair (e.g. 10 mg of prednisone used for replacement therapy for adrenal insufficiency)
* Patients who are lactating
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; and cirrhosis. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection (except for uncomplicated urinary tract infection), interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have received any of the prohibited medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
3 year recurrence-free survival | Time from study entry (randomization) to the time of cancer recurrence, assessed at 3 years
  Will be estimated using the Kaplan Meier method and treatment comparisons will be made using a stratified log-rank test.

SECONDARY OUTCOMES:
Incidence of adverse events | 12 months
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) by treatment regimen. Will be evaluated descriptively using frequencies and percentages and will be reported using tables. Differences between treatment arms will be assessed through absolute deviations and contingency table analyses. All patients who receive treatment, will be evaluated for toxicity. Toxicities by type and maximum grade over the course of treatment and follow up will be summarized and by date of occurrence (acute toxicity and late adverse effects).
Recurrence patterns | 5 years
  The cumulative incidences of vaginal recurrence, pelvic recurrence, retroperitoneal, and distant recurrence from endometrial cancer will be estimated within treatment regimen. Treatments will be compared graphically using Kaplan-Meier estimates of the survival function.
5 year recurrence free survival | Time from study entry (randomization) to the time of cancer recurrence, assessed at 5 years
  Proportions will be compared by treatment using Fisher's exact test. This analysis may be delayed until the data are mature.
Overall survival | Duration of time from study entry to time of death or the date of last contact, assessed up to 5 years
  Will be estimated using the Kaplan Meier method and treatment comparisons will be made using a stratified log-rank test.
Patient-reported outcomes | Up to 2 years after starting treatment
  Will be assessed by questionnaire.
Impact of circulating tumor deoxyribonucleic acid (ctDNA) on treatment outcomes | Up to 5 years
  Will examine the association between ctDNA and 2- year (or 3-year) progression free survival in a 2-stages of analysis.

OTHER OUTCOMES:
Potential transformations of the severity of adverse events | 12 months
  An example of potential transformation of the severity of adverse events is whether or not the patient experienced >= grade 3 events. It will be assessed by CTCAE and treatment regimen.
Biomarker analysis | Baseline
  Will assess baseline genetic characteristics (e.g. mutations) and microenvironment parameters, treatment, and interactions between treatment and biomarkers in a Cox regression.
Functional Assessment of Cancer Therapy (FACT)-Immune Checkpoint Modulator (ICM) subscale | Up to 2 years after starting treatment
  Treatment differences in the FACT-ICM subscale and self-reported bother from side effects will be explored using a linear mixed model for repeated measures, adjusted for the baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Floor Backes, Principal Investigator — NRG Oncology
Locations (280):
- United States (275):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - GenesisCare USA - FGO, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (5):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692
- [Derived] Liu YL, Stadler ZK. The Future of Parallel Tumor and Germline Genetic Testing: Is There a Role for All Patients With Cancer? J Natl Compr Canc Netw. 2021 Jul 28;19(7):871-878. doi: 10.6004/jnccn.2021.7044. PMID 34340209

DOCUMENTS (1):
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT04214067/ICF_000.pdf